CLINICAL TRIAL: NCT03132857
Title: The State of Play in Picardy of the Knowledge of the Elderly at Risk of Falling at Home in Terms of Prevention and Evaluation.
Acronym: Epic-SaPE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: RNI2016-39 Dr Moyet
Record Dates: First submitted 2017-04-14; First posted 2017-04-28 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Knowledge, Attitudes, Practice; Elderly
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assess the state of knowledge of the subjects falling or at risk, their risk of recurrence or first episode, compared to medical knowledge. — Assess the state of knowledge of the subjects falling or at risk, their risk of recurrence or first episode, compared to medical knowledge.

SUMMARY:
In 2010, the French population over 75 years of age was 9%; It will be 13% in 2030 and 19% in 2050 according to estimates. The incidence of falls is high in the elderly population, with at least one fall per year for one-third of the over-65s and for half of the over-80s. These data are consistent with the international medical literature, particularly in Japan, the United States and France, with a high rate of recurrence from the first fall. Falling is a complex phenomenon that is of great importance in terms of morbidity and mortality since it can be followed by serious complications: failure to recover, recurrences, trauma (fractures, hematomas, wounds), complications of decubitus and ulcers, Immobilization, loss of autonomy, hospitalization, institutionalization, psychological complications (post-fall syndrome, depressive syndrome), death.

Fall risk factors are well known and described and relayed by learned societies of geriatrics and medical literature. In addition, HAS reported on this issue in 2009.

The French Society of Geriatrics and Gerontology (SFGG) defines fragility as a clinical syndrome that reflects a decrease in reserve physiological capacities that alters the coping mechanisms of stress. Its clinical expression is modulated by comorbidities and psychological, social, economic and behavioral factors. Frailty syndrome is a risk marker for mortality and pejorative events, including disability, falls, hospitalization and institutionalization. The fall and its complications are closely related to the fragility syndrome. The very fragile patient must take an active part in his own care. He is the first advocate of fall prevention.

On the other hand medical desertification and the low number of geriatricians makes this implication problematic even more so if the person is isolated or has cognitive impairment. Nevertheless, it is important to make the patient actor of his own prevention. This is the first study to describe the knowledge of older adults about their own risk of falling.

ELIGIBILITY:
Inclusion Criteria:

* male or female over 75
* considered by their attending physician as a fall arrester or at risk of falling and living at home
* presenting themselves to the office of their attending physician for a consultation for whatever reason.

Exclusion Criteria:

* EHPAD resident
* patient not affiliated to a social security scheme
* under legal protection

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly Picard subjects, living at home in fall risk factor and assessing their own risk of falling.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2017-03-12 (Actual); Primary Completion 2017-12-16 (Actual); Study Completion 2017-12-16 (Actual)

PRIMARY OUTCOMES:
Analysis of a closed-response questionnaire on the risk of falling older adults. | 1 day
  Questionnaire with closed answers, based on the recommendations of the HAS (high authority of health) 2009 and the recommendations of the SFGG (French Society of Geriatrics and Gerontology) concerning the risk of fall of the elderly subject.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France